CLINICAL TRIAL: NCT02044328
Title: Icotinib as an Adjuvant Therapy for Patients With Stage IIA-IIIA Adenocarcinoma With EGFR Mutation: a Prospective, Exploratory Study
Brief Title: Icotinib as an Adjuvant Therapy for Patients With Stage IIA-IIIA Adenocarcinoma With EGFR Mutation
Acronym: ICAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV57
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib (Experimental): Patients receive icotinib 125 mg three times daily as adjuvant chemotherapy with for 18 months after surgery.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib is administered 125 mg three times per day.
  Other Names: Commana; BPI-2009

SUMMARY:
Adjuvant therapy has been proved effective in treating earlier stage or less advanced non-small-cell lung cancer. This study is designed to evaluate the efficacy of icotinib as adjuvant therapy in treating stage IIA-IIIA adenocarcinoma patients with EGFR mutation. The primary endpoint is disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* The patients present with operable stage IIA-IIIA (N0-1) lung adenocarcinoma with 19 or 21 exon mutation
* The patients have no history of anti-cancer therapies including chemotherapy, radiation therapy
* The patients' Eastern Cooperative Oncology Group scores are ≤ 0-1
* The patients signed the written informed consent

Exclusion Criteria:

* Patients with unresected tumor
* Wild EGFR type
* Allergic to the study drug
* Patients have severe non-cancerous diseases
* Patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years

SECONDARY OUTCOMES:
1-year Survival Rates | 1 year
3-year Survival Rates | 3 years
Number of patients suffered adverse events | 42 months
  Adverse events are evaluated and coded by Common Terminology Criteria for Adverse Events version 4.0

OTHER OUTCOMES:
Difference of disease-free survival by status of Bcl-2 interacting mediator of cell death | 2 years
  Compare the disease-free survival between patients with positive Bcl-2 interacting mediator of cell death mutation and patients without this mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yi, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China